CLINICAL TRIAL: NCT06342583
Title: Advanced Social Relations Training for Children and Young People With Autism Spectrum Disorder
Brief Title: Advanced Social Relations Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2024-004
Record Dates: First submitted 2024-03-11; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; children; social relation; awareness on social media; communication; social stories
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 15 children from the experimental group will see social stories on a technological device (PC, tablet) and then see slides on a technological device concerning the correct use of social media.
  Interventions: Other: Advanced social relations training with technical device
- Traditional group (Other): 15 children in the control group will see social stories in paper form (flashcards) and then be exposed to the explanation of risks and correct use of social media in a traditional way (flashcards).
  Interventions: Other: Advanced social relations training without technical device

INTERVENTIONS:
Other: Advanced social relations training with technical device — 15 participants from the experimental group will undergo a first part in which they will be guided through social stories to construct an appropriate conversation repertoire. In the first phase the participants will see 8 social stories with scenes from everyday life and after learning the correct mode of interaction and communication they will be asked to interact in the group by playing the roles previously seen in the social stories. These will be shown on a technological device. Participants will have the opportunity to choose the correct mode of interaction by selecting it directly on the technological device. Each selected alternative will refer to the next scenario in relation to the selected answers. In the second phase participants will be instructed on the correct use of social media. Slides will be shown to explain risks and correct use and the operator will show on the technological device (Smartphone) all the practical steps to be taken (e.g. privacy settings).
  Arms: Experimental group
Other: Advanced social relations training without technical device — 15 participants from the control group will undergo a first part in which they will be guided through social stories to build an appropriate conversation repertoire. In the first phase, the participants will see eight social stories illustrating scenes from everyday life and, after learning the correct modes of interaction and communication, they will be invited to interact in the group by playing the roles previously seen in the social stories. These will be shown in traditional mode (flashcards). Participants will have the opportunity to choose the correct mode of interaction by touching the card showing the appropriate mode. Each selected alternative will refer to the next scenario in relation to the selected answers. In the second phase participants will be instructed on the correct use of social media (facebook, instagram, TikTok, Whatsapp, YouTube). The trainer will show images on paper related to risks and correct use of social media.
  Arms: Traditional group

SUMMARY:
Advanced social relations protocol is aimed at young people with autism aged 9-12 years with an intelligence quotient (IQ) ≥ 80. There will be an experimental group in which technology will be used and a control group in which activities will be carried out in the traditional way. The protocol will be carried out once a week for a duration of 45 minutes. The aim is to enhance communication and social skills within the group. A total of 23 sessions are planned. From the first to the third session the participants will acquire skills for communicating and conversing in an appropriate way. Thereafter from the fourth to the eleventh session social stories illustrating scenes from everyday life will be shown, with the aim of learning and managing the dynamics in which they find themselves on a daily basis. At the end of each story shown they will be asked to impersonate the protagonists depicted in the stories, each participant involved in turn will play all the roles shown in the stories, thus working in the mode of role playing.

The last part, which includes sessions from the twelfth to the twenty-third, will be dedicated to the correct and conscious use of social networks with a focus on the risks that can be encountered and the correct ways to make good use of them.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of autism
* intelligence quotient ≥ 80

Exclusion Criteria:

* presence of other medical disorders

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-17 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Vineland-II (Vineland Adaptive Behavior Scales-II - Survey Intervention Form) | the administration of the Vineland-II takes approximately 20-60 minutes
  The Vineland-II, a revision of the Vineland Adaptive Behavior Scales (Vineland ABS), assess adaptive behavior (AB), i.e., the activities that the individual habitually performs to meet the expectations of personal autonomy and social responsibility characteristic of people of the same age and cultural background.
  Specifically, they aim to measure AB in the domains Communication, Skills of Daily Living, Socialization (in individuals from 0 to 90 years of age) and Motor Skills (in individuals from 0 to 7 years of age and 56 to 90 years of age). Assessment of AB is necessary for diagnosis of intellectual disability disorder and, in accordance with Diagnostic and Statistical Manual of Mental Disorders (DSM-5), for assessment of the level of severity of the disorder.
  The Vineland-IIs consist of 4 scales divided into 11 subscales. They also provide an overall AB index.
Eye contact | the administration of the test takes approximately 10 minutes
  Unit of measurement: Number of visual contacts observed during social interaction.
  Rating scale: 0 to 10, where 0 indicates no eye contact and 10 indicates constant eye contact
Smile in relation to group members' expressions | the administration of the test takes approximately 10 minutes
  Unit of measurement: Number of smiles observed in relation to group members' expressions.
  Rating scale: 0 to 10, where 0 represents no smiles and 10 indicates constant smiling in response to others' expression Unit of measurement: Number of greetings performed during social interaction. Rating scale: 0 to 10, where 0 indicates absence of greetings and 10 indicates a high number of greetings
Greeting | the administration of the test takes approximately 10 minutes
  Unit of measurement: Number of greetings performed during social interaction. Rating scale: 0 to 10, where 0 indicates absence of greetings and 10 indicates a high number of greetings
Asking a question | the administration of the test takes approximately 10 minutes
  Unit of measurement: Number of questions asked during social interaction. Rating scale: 0 to 10, where 0 indicates no questions and 10 indicates a high number of questions
Proposing an idea or activity to be carried out | the administration of the test takes approximately 10 minutes
  Unit of measurement: Number of ideas or activities proposed during social interaction.
  Rating scale: 0 to 10, where 0 indicates no proposals and 10 indicates a high number of proposals
Answering a question | the administration of the test takes approximately 10 minutes
  Unit of measurement: Percentage of questions answered during social interaction. Rating scale: From 0% (no response) to 100% (response to all questions)
Taking verbal initiative | the administration of the test takes approximately 10 minutes
  Unit of measurement: Number of times verbal initiative is taken during social interaction.
  Rating scale: 0 to 10, where 0 indicates no verbal initiative and 10 indicates high verbal initiative
Approval/sharing gestures | the administration of the test takes approximately 10 minutes
  Unit of measurement: Number of approval or sharing gestures observed during social interaction.
  Rating scale: 0 to 10, where 0 indicates no approval/sharing gestures and 10 indicates a high frequency of such gestures.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Istituto per la Ricerca e l'Innovazione Biomedica
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ALMUMEN, H., & ALMUHAREB, K. (n.d.). Intervento di storia sociale arricchita dalla tecnologia: coinvolgere i bambini con disturbi dello spettro autistico nella comunicazione sociale. International Journal of Early Childhood Special Education, 12(1), 96-119. https://doi.org/10.20489/intjecse.726397
- [Background] Camilleri LJ, Maras K, Brosnan M. The impact of using digitally-mediated social stories on the perceived competence and attitudes of parents and practitioners supporting children with autism. PLoS One. 2022 Jan 18;17(1):e0262598. doi: 10.1371/journal.pone.0262598. eCollection 2022. PMID 35041714